CLINICAL TRIAL: NCT01183377
Title: Screening of Menstrual Disorder in Elite Feamle Athlete in Iran
Brief Title: Frequency of Female Athlete Triad Among Elite Female Athlete of Iran in Different Sport in 2007
Status: Terminated | Type: Observational
Why Stopped: the study terminated last week
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Rheumatology Research Center, Haleh Dadgostar
Other Study IDs: 85-01-41-3488
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Menstruation Disturbances; Eating Disorder; Bone Loss
Keywords: Female Athlete Triad syndrom; Eating disorder; osteoprosis
MeSH Terms: conditions — Menstruation Disturbances; Feeding and Eating Disorders; Bone Diseases, Metabolic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Female athlete Triad syndrom was based on menstrual disorder,Eating Disorder and bone loss

SUMMARY:
Women's evermore presence in professional and athletic sports has revealed sound evidence on the existence of female athlete triad among the world's elite female athletes. This triad consists of eating disorders, amenorrhea and osteoporosis. It has been stated that all female athletes are potentially at risk, but it is not clear to what extent those exercising at different levels are at risk of this syndrome/triad. Since the manifestation of this triad is often denied, or under-reported, appropriate screening methods are required to identify the symptoms. There is still no clear-cut information available on the incidence of this triad in Iran. And there are religious and cultural differences between Iran's elite female athletes and those in other countries. Therefore, in order to meet Iranian female athletes' needs, the investigators decided to determine the frequency of the female athlete triad in Iran.

ELIGIBILITY:
Inclusion Criteria:

* All Elite Female athletes who play in international teams in sport federation or champion Team in Tehran between 13-45 years old.

Exclusion Criteria:

* The 13-15 year old female athletes who are not manarch with secondary sex charactristics.

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population: Professional Iranian female athletes who are members in national teams or federations sports and champion team in Tehran
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Female Athlete Triad among Elite female athlete in Iran in 2006 | 24 month

SECONDARY OUTCOMES:
prevalence of menstrual disorder in female athlete in Iran in 2006 | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Haleh Dadgostar, MD, Study Director — Rheumatology Research Center, Tehran University for Medical Sciences; Fereydoun Davatchi, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Shafie Movaseghi, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; ashraf Aleyasin, MD, Principal Investigator — Tehran University for Medical Sciences; mohamad hosein Forozanfar, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Talia Alenabi, MD, Principal Investigator — Sport Medicine Federation of Islamic Republic Of Iran; Narges Chime, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; pooneh Kimia ghalam, MD, Principal Investigator — Health ministry of Iran
Locations (1):
- Rheumatology Research Center, Shariati Hospital, Tehran, Tehran Province, Iran